CLINICAL TRIAL: NCT06320496
Title: Evaluation of the Effect of a Physical Activity Recovery Stay on the Physical Condition and Quality of Life of Children in a Situation of Physical Deconditioning
Brief Title: Evaluation of the Effect of a Physical Activity Recovery Stay
Status: Recruiting | Type: Observational
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Other Study IDs: IRR-FLAVIGNY-2021-2
Record Dates: First submitted 2024-02-05; First posted 2024-03-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Children With Cerebral Palsy; Children With Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Deconditioning to physical exertion: The children taking part in the return-to-physical-activity program are referred to the Flavigny-sur-Moselle CMPRE for medical consultation due to a state of deconditioning to physical exertion concomitant with a pathological situation. The pathology most frequently encountered during this stay is cerebral palsy. However, the Flavigny CMPRE is accredited in a number of fields (orthopedics, burns, neurology, oncology), and the pathologies of the children referred to this stay are representative of these. These include children with scoliosis, obesity, Guillain-Barré syndrome, cystic fibrosis, Charcot's disease and cancer.

SUMMARY:
A WHO study in 2020 revealed that 81% of adolescents (aged 11-17) do not respect the recommendation of one hour of moderate physical activity per day. In the context of disability, many factors impose limits on physical activity. While the pathology itself induces limitations and restrictions (prolonged sitting time, assisted movement, etc.), organizational constraints also apply to both children and parents, who have to divide their time between work, school and therapeutic care, which is sometimes numerous and varied over the course of a single week. These limitations generate stress and fatigue, and prolonged sedentary periods lead children with chronic illnesses, rare diseases or disabilities into a process of physical deconditioning. The accumulation of sedentary time is detrimental to cardiovascular and metabolic health.

To combat this deconditioning, the 2008 National Physical Activity and Sport Plan (PNAPS) sets out the main guidelines for treatment and implementation. The plan explains that "for patients with chronic illnesses, rare diseases or disabilities, the aim is to encourage care and guidance towards Adapted Physical Activity (APA). The attending physician will be able to identify local therapeutic education programs, rehabilitation services and "sport-santé" offers, to improve access for these patients to supervised local programs". In addition, the plan suggests "developing APA programs in healthcare establishments to enable people with chronic illnesses, rare diseases or disabilities to access health education incorporating practical sessions".

In line with this plan, an exercise reconditioning program has been set up at our facility. This three-month stay includes children with a variety of pathologies, but with a common feature of physical deconditioning.

ELIGIBILITY:
Inclusion Criteria:

* Children with a pathology (chronic disease, rare disease or disability) in a state of deconditioning to exercise
* Taken in charge at the CMPRE for a stay to resume physical activity

Exclusion Criteria:

* Age under 8 and over 18
* Patients undergoing rehabilitation during the stay
* Patients with a significant change in their therapeutic management during the stay
* Significant cognitive impairment preventing comprehension of instructions
* Significant club or leisure sports activity (3x/week)
* Electric wheelchair
* Non-compliance with stay (5 ½ days missed out of total stay)
* Participation in another study during the return-to-physical-activity stay

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The children taking part in the return-to-physical-activity program are referred to the Flavigny-sur-Moselle CMPRE for medical consultation due to a state of deconditioning to physical exertion concomitant with a pathological situation. The pathology most frequently encountered during this stay is cerebral palsy. However, the Flavigny CMPRE is accredited in a number of fields (orthopedics, burns, neurology, oncology), and the pathologies of the children referred to this stay are representative of these. These include children with scoliosis, obesity, Guillain-Barré syndrome, cystic fibrosis, Charcot's disease and cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnoform test score | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  To evaluate the effect of the return to physical activity stay prescribed by the doctors at the Flavigny CMPRE on the physical condition of the children taking part in the stay Score between 0 and 20 for each part of the test, with 20 being the best score (and therefore the best physical condition).

SECONDARY OUTCOMES:
KidScreen52 quality-of-life scale score. | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Quality of life scale : a T-score value is calculated. Scores range from 10 to 50, where 10 represents the lowest possible value and thus a very low health-related quality of life and 50 the maximum value, i.e. a very high health-related quality of life.
Impedance measurement | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Recording weight on a balance : Ideally, the patient should have lost weight by the end of the reconditioning stay.
Exercise test on ergometer | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Three-minute warm-up without resistance, then increase in difficulty every minute until you reach 80% of your theoretical maximum heart rate.
Anamnesis | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  description of the antecedents
6-minute walk test | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Walk the maximum distance for 6 minutes
Energy expenditure index | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Functional walking index calculated during a regular, spontaneous 5-minute walk. This index is equal to the ratio of heart rate averaged over the 5th minute to walking speed.
Gluteal bridge | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Physical exercise that helps to strengthen the gluteus muscles (located in the buttocks) and hamstrings. The longer you hold the position, the better is.
Shirado test | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Assessment of abdominal endurance: keep your shoulders off the ground while lying on your back with your feet raised. The maximum duration of this test is three minutes. Low performance if time less than 60 seconds, maximum if time greater than 150 seconds.
Sorensen test | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Assessment of trunk extensor endurance: hold the weight of your trunk in isometric position for as long as possible, with your arms crossed over your chest. The maximum duration of this test is 240 seconds. The longer the position is maintained, the better.
Timed Up and Down Stairs (TUDS) test | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  he participant stands 1 foot from the bottom of a 14-step flight of stairs. The participant is instructed to "Quickly, but safely go up the stairs, turn around on the top step (landing) and come all the way down until both feet land on the bottom step (landing." The participants are allowed to choose any method of traversing the stairs. The TUDS score was the time in seconds from the "go" cue until the second foot returned to the bottom landing. Shorter times indicated better functional ability.
Floor survey test | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Evaluation and exercise element designed to teach the subject to get up from the ground using the righting sequence
Mini Bestest : Each of the 14 tests is graded from 0 to 2. "0" represents the lowest functional level and "2" the highest functional level. Maximal score : 28. | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Clinical assessment of postural control
The Canadian Occupational Performance Measure | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  Tool used in occupational therapy to identify people's occupational problems
A motivational questionnaire | Day of patient inclusion and 3 months after, day on which the study ends for the patient
  A tool for assessing involvement and motivation levels : 7 questions score between 0 and 10. 0 = no motivation 10 = total motivation

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France

IPD SHARING:
Plan to Share IPD: No